CLINICAL TRIAL: NCT03825432
Title: Investigation of Physical Activity and Associated Factors in Lower Extremity Amputees
Status: Completed | Type: Observational
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Sponsor
Other Study IDs: ETK00-2018-0068
Record Dates: First submitted 2019-01-24; First posted 2019-01-31 (Actual); Last update posted 2021-10-14 (Actual); Status verified 2021-10

CONDITIONS: Amputee
Keywords: Physical activity; Prosthesis
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study was to investigate the physical activity and related factors of individuals with lower extremity amputation.

Participants in the study who have signed a voluntary consent form will be informed about the study first.Then, demographic information form will be started to be recorded in order to inform the socio-demographic characteristics of the participants and the information about amputation and prosthesis. The participants will be given the Timed Up and Go Test, L Test, Functional Reach Test and 2 Minute Walk Test. Following these tests, participants will continue with the scales to be answered by the participants themselves.These are respectively; Activity-Specific Balance Confidence Scale, Trinity Amputation and Prosthesis Experience Scale and Amputee Body Image Scale.Before the data is collected, individuals will be informed about the equipment to be used in the tests.An adequate number of trials will be conducted before the evaluation and use of the equipment in order to be familiar with the equipment. All assessments will be made by the same physiotherapist.

DETAILED DESCRIPTION:
Amputation affects the quality of life of the individual; It is an important surgical intervention that can lead to functional, psychological and social isolation. The prevalence and incidence of amputation is difficult to determine precisely at the international level.The etiology of amputation varies depending on geographical location.Peripheral vascular diseases are the most common causes of amputation in developed countries and trauma in developing countries.Limitations in body composition and function after amputation decrease the activity level, so the participation of amputees is negatively affected.Physical activity refers to any activity involving body movement and increasing the heart rate and respiratory rate of the individual.

Most of the lower extremity amputated patients had low levels of physical activity and participation in sports activities; It was also found that individuals with lower extremity amputations were less active than those without lower extremity amputation.However, there are few studies that have shown that individuals with lower extremity amputation are regularly active, and the amputation of amputated individuals in these studies has mostly caused traumatic amputations.

Lower extremity amputation; Although there is significant evidence showing that the risk of developing a number of chronic degenerative diseases such as cardiovascular disease, diabetes, hypertension, obesity and osteoarthritis significantly increases, there are few studies investigating and investigating physical activity after amputation.Despite these investigations, relatively little is known about the components or models of physical activity necessary to provide protection against chronic diseases and to improve metabolic health in these specific population groups. Therefore, accurate measurement and estimation of the level of physical activity and energy expenditure is critical in the prevention and prevention of chronic diseases in individuals with lower extremity amputation.

A higher level of physical activity is associated with better perceived quality of life in individuals with lower extremity amputation.Therefore, it is important to develop physical activity in individuals with lower extremity amputations.

Although there are studies investigating the physical activity in individuals with lower extremity amputation as a result of our literature review, no study has been found investigating factors related to physical activity.

The aim of this study was to investigate the physical activity and related factors of individuals with lower extremity amputation.

RESEARCH QUESTIONS

Question 1: What is the level of physical activity in individuals with lower extremity amputation?

Question 2: What are the factors associated with the level of physical activity in amputees of the lower extremity?

THE UNIVERSE AND THE SAMPLING OF RESEARCH

The individuals to be included in the study will be selected from voluntary amputees who apply to the Prosthesis-Orthotics Biomechanics Unit of the Department of Physiotherapy and Rehabilitation of the Eastern Mediterranean University Faculty of Health Sciences.

As the sample volume in the study was to be linear regression analysis by using G-Power program, it was determined that the total determinant factor number would be 8 and 108 people as alpha, 0.05, beta: 0.80 and effect size as 0.15.

METHOD OF RESEARCH

Participants in the study who have signed a voluntary consent form will be informed about the study first.Then, demographic information form will be started to be recorded in order to inform the socio-demographic characteristics of the participants and the information about amputation and prosthesis.The participants will be given the Timed Up and Go Test, L Test, Functional Reach Test and 2 Minute Walk Test. Following these tests, participants will continue with the scales to be answered by the participants themselves.These are respectively; Activity-Specific Balance Confidence Scale, Trinity Amputation and Prosthesis Experience Scale and Amputee Body Image Scale.Before the data is collected, individuals will be informed about the equipment to be used in the tests.An adequate number of trials will be conducted before the evaluation and use of the equipment in order to be familiar with the equipment. All assessments will be made by the same physiotherapist.

INCLUDING CRITERIA

* Use prosthesis for at least 6 months
* 18 years to 85 years
* Independent walking distance of 30 meters
* Individuals with unilateral amputation will be included.

EVALUATIONS IN THE RESEARCH

In this study, age, gender, height, body weight, body mass index, educational status, marital status, profession, socio-demographic characteristics of the dominant side, as well as the history of amputation, cause of amputation, amputation side and level, stump shape, phantom pain Factors related to amputation, such as phantom sensation, type of prosthesis and duration of use will be recorded with the form prepared.

Timed Up and Go Test: Timed Up and Go Test will be used to measure the risk of functional mobility and fall.The participant seated on the chair without clinging to his arms 3m from the ground, 3m after walking without touching a place to return, the chair will be asked to go back to the sitting position and the time will be recorded in seconds..

L Test: The L test will be used to assess functional mobility. In the L-shaped direction, the participants will be carried out on the ground where the long edge of L is 7 meters and the short edge will be 3 meters. At the beginning of the test, the participants will sit in a chair without arms and stand up from the chair with the start command, complete the L shape at the preferred speed and return to the chair without interruption. Thus, a total distance of 20 meters will be completed at the end of the test. The completion time of the test will be recorded.The intrarater reliability of the test was found to be 0.97 and the interrater reliability was 0.96, and it was shown to have a very high validity.

Functional Reach Test: The Functional Reach Test will be done to evaluate the stability limits and fall risks of individuals.For the test, individuals will be asked to stand upright on their shoulders with their shoulders wide open.In this position, the acromion level of individuals will be marked on the wall.Individuals will be asked to lift their arms forward to the marked level and to reach forwards without moving their feet.The distance between the start and end position will be measured and recorded in cm.The test will be repeated 3 times and the measurements will be averaged.The test will be repeated if individuals touch the wall or take steps during the test.

2-Minute Walk Test: 2 Minute Walk Test will be used to evaluate the functional capacity of individuals.The patient will be seated in the chair at the 25-meter track where the test will be done and the distance within 2 minutes will be measured in meters.Before and after the test, the patient's pulse and oxygen saturation with pulse oximetry will be measured and recorded using the Borg Scale.

Activity-Specific Balance Confidence Scale: In order to evaluate the reliability of the balance, the Activity-Specific Balance Confidence Scale, which has been validated for Turkish reliability and validity, will be used.There are 16 functional activities in the scale. Each individual will have 16 different activities and the reliability will be evaluated accordingly.Measurement results from 0% to 100% are given.0% ir 'no trust' 'and 100% 100' completely sure ''.If this scale gives a score above 80%, then it is mentioned that the balance is reliable.For internal consistency, the Cronbach's alpha value was 0.9649 for the test and 0.9648 for the retest.

Trinity Amputation and Prosthesis Experience Scale: In order to evaluate the quality of life, the Trinity Amputation and Prosthesis Experience Scale which is a validity and validity scale in amputees will be used. Trinity Amputation and Prosthesis Experience Scale two consists of parts.In the first part; psychosocial adjustment, activity restriction and prosthesis satisfaction.In the second part; questions about how many hours the prosthesis is worn, general health and physical capacity. For internal consistency, Cronbach's alpha value for psychosocial adjustment; 0.862 for activity restriction; 0.894 and 0.915 for prosthetic satisfaction.

Amputated Body Image Scale: The Amputee Body Image Scale, which has been validated for Turkish validity and reliability, will be used to assess body image disorders in amputees. This 20-item scale evaluates the situations that the amputee perceives and feels about the body. The score obtained varies between 20-100. A high score indicates a poor body image. The Cronbach alpha value was 0.939.

Assessment of Physical Activity: Sociodemographic data such as age, height, weight and gender from subjects will be recorded on the accelerometer profile using Stay Healthy software (Research Tracker 6, Version 3.1, Stay Healthy, Inc., Monrovia, USA). The data will be collected in computer environment as total calorie and efficiency count (VM; X axis, Y axis, Z axis).The total calories will be recorded in kilocalories, while the data count will be recorded in terms of acceleration.

ELIGIBILITY:
Inclusion Criteria:

* Use prosthesis for at least 6 months
* 18 years to 85 years old subjects
* Independent walking distance of 30 meters
* Individuals with unilateral amputation will be included

Exclusion Criteria

• Bilateral amputees

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Lower Limb Amputees
Sampling Method: Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2019-02-20 (Actual); Primary Completion 2019-07-16 (Actual); Study Completion 2019-07-16 (Actual)

PRIMARY OUTCOMES:
Physical activity | 3 days
  Physical activity of the subjects will be recorded by an accelerometer (Research Tracker 6, Version 3.1, Stay Healthy, Inc., Monrovia, USA) in kilocalories.

SECONDARY OUTCOMES:
Timed Up and Go Test | The test will be performed in the first day of assessment of each amputee for once after enrollment. It takes about 5 minutes.
  Timed Up and Go Test will be used to measure the risk of functional mobility and fall. The participant seated on the chair without clinging to his arms 3m from the ground, 3m after walking without touching a place to return, the chair will be asked to go back to the sitting position and the time will be recorded in seconds. Shorter time means better mobility function.
L Test | The test will be performed in the first day of assessment of each amputee for once after enrollment. It takes about 5 minutes.
  The L test will be used to assess functional mobility. In the L-shaped direction, the participants will be carried out on the ground where the long edge of L is 7 meters and the short edge will be 3 meters. At the beginning of the test, the participants will sit in a chair without arms and stand up from the chair with the start command, complete the L shape at the preferred speed and return to the chair without interruption. Thus, a total distance of 20 meters will be completed at the end of the test. The time will be recorded in seconds that shorter time means better mobility function.
Functional Reach Test | The test will be performed in the first day of assessment of each amputee for once after enrollment. It takes about 2 minutes.
  The Functional Reach Test will be done to evaluate the stability limits and fall risks of individuals. For the test, individuals will be asked to stand upright on their shoulders with their shoulders wide open. In this position, the acromion level of individuals will be marked on the wall. Individuals will be asked to lift their arms forward to the marked level and to reach forwards without moving their feet. The distance between the start and end position will be measured and recorded in cm that higher distance means better balance.
2 Minute Walk Test | The test will be performed in the first day of assessment of each amputee for once after enrollment. It takes about 3 minutes.
  2 Minute Walk Test will be used to evaluate the functional capacity of individuals. The patient will be seated in the chair at the 25-meter track where the test will be done and the distance within 2 minutes will be measured in meters. Longer distance means better ambulation capacity.
Activities-Specific Balance Confidence Scale | The scale will be performed in the first day of assessment of each amputee for once after enrollment. It takes about 2 minutes.
  In order to evaluate the reliability of the balance, the Activity-Specific Balance Confidence Scale, which has been validated for Turkish reliability and validity, will be used. There are 16 functional activities in the scale. Each individual will have 16 different activities and the reliability will be evaluated accordingly.Measurement results from 0% to 100% are given.0% 'no trust' 'and 100% 100' completely sure ''. The higher score means better balance confidence.
Amputee Body Image Scale | The scale will be performed in the first day of assessment of each amputee for once after enrollment. It takes about 2 minutes.
  The Amputee Body Image Scale, which has been validated for Turkish validity and reliability, will be used to assess body image disorders in amputees. This 20-item scale evaluates the situations that the amputee perceives and feels about the body. The score obtained varies between 20-100. The higher score indicates worse body image.
Trinity Amputation and Prosthesis Experience Scale, Psychosocial adjustment subscale | The scale will be performed in the first day of assessment of each amputee for once after enrollment. It takes about 3 minutes.
  In order to evaluate psychosocial condition, psychosocial adjustment subscale of the Trinity Amputation and Prosthesis Experience Scale scores between 5-25 that higher means better psychosocial condition.
Trinity Amputation and Prosthesis Experience Scale, Activity restriction subscale | The scale will be performed in the first day of assessment of each amputee for once after enrollment. It takes about 3 minutes.
  In order to evaluate activity restriction, activity restriction subscale of the Trinity Amputation and Prosthesis Experience Scale scores between 4-12 that higher means higher activity restriction.
Trinity Amputation and Prosthesis Experience Scale, Prosthesis satisfaction subscale | The scale will be performed in the first day of assessment of each amputee for once after enrollment. It takes about 3 minutes.
  In order to evaluate prosthesis satisfaction, prosthesis satisfaction subscale of the Trinity Amputation and Prosthesis Experience Scale scores between 10-50 that higher means better prosthetic satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Yasin YURT, Asst.Prof., Study Director — Eastern Mediterranean University
Locations (1):
- Eastern Mediterranean University, Mersin, Turkey (Türkiye)